CLINICAL TRIAL: NCT06844474
Title: A Phase II, Multicenter, Open-Label Clinical Study to Evaluate the Safety, Tolerability and Efficacy of SHR-1826 for Injection in Patients With NSCLC
Brief Title: A Phase II Clinical Study of SHR-1826 for Injection in Patients With NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1826-203
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): SHR-1826 for injection in combination with Adebrelimab injection and SHR-8068 with or without Bevacizumab injection
  Interventions: Drug: SHR-1826；Adebrelimab；SHR-8068；Bevacizumab

INTERVENTIONS:
Drug: SHR-1826；Adebrelimab；SHR-8068；Bevacizumab — Drug:
  Drug: SHR-1826 Administration by intravenous infusion for a cycle of 3 weeks.
  Drug: Adebrelimab Administration by intravenous infusion for a cycle of 3 weeks.
  Drug: SHR-8068 Administration by intravenous infusion for a cycle of 6 weeks.
  Drug: Bevacizumab Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This study is an open-label, multicenter Phase II clinical trial to evaluate the safety, tolerability and efficacy of SHR-1826 for injection in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. ECOG performance score of 0-1.
3. Life expectancy ≥ 3 months.
4. Have at least one measurable tumor lesion per RECIST v1.1.
5. Subjects with histologically confirmed locally advanced or metastatic NSCLC.
6. Good level of organ function.
7. Provide archived or fresh tumor tissue for vendor test.

Exclusion Criteria:

1. Subjects with active central nervous system metastases or meningeal metastases;
2. History of serious cardiovascular and cerebrovascular diseases;
3. Subjects with a history of interstitial pneumonitis or imaging at screening suggestive of suspected interstitial pneumonitis;
4. Severe infection within 4 weeks prior to the first dose;
5. Ongoing or previous anti-tumor therapies within 4 weeks prior to the first dose of study drug;
6. Subjects with uncontrolled tumor-related pain;
7. Received >30 Gy of non-thoracic radical radiation therapy within 4 weeks prior to the first administration of study drug;
8. Concomitant other malignancies ≤ 5 years prior to first dose of study drug;
9. Unresolved toxicities from previous anti-tumor therapy to ≤ Grade 1 (based on NCI CTCAE v5.0);
10. History of immunodeficiency, including a positive HIV test;
11. Per the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) /serious adverse events(SAEs) | approximately 2 years
Overall response rate (ORR) | approximately to 2 years

SECONDARY OUTCOMES:
Duration of response (DoR) | approximately to 2 years
Disease control rate (DCR) | approximately to 2 years
Progression-free survival (PFS) | approximately to 2 years
Overall survival (OS) | approximately to 5 years after last subject enrolled

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army (PLA) General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided